CLINICAL TRIAL: NCT06960408
Title: Effects of Sleep Hygiene Education and Progressive Relaxation Exercise on Anxiety, Sleep Quality and Glycemic Control in Type 2 Diabetic Patients: A Randomized Controlled Trial
Brief Title: Effects of Sleep Hygiene Education and Progressive Relaxation Exercise on Anxiety, Sleep Quality and Glycemic Control in Diabetic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ülkü Görgülü Polat, Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2285360200
Record Dates: First submitted 2025-04-07; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: sleep; type 2 diabetes mellitus; Progressive muscle relaxation; Sleep quality; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: intervention group (Experimental): The study will be conducted with diabetic individuals who come to the endocrine clinic. The study will be conducted for 6 months. Intervention group Individuals who accept the study will be given face-to-face Progressive Relaxation Exercise training by the researcher in the first week of the first month of the study and will be applied. The Progressive Relaxation Exercise application will also be sent to the patient via WhatsApp and will be applied with the researcher via online interviews in the 2nd, 3rd and 4th weeks for 30 minutes 3 days a week (Monday-Wednesday-Friday). From the 2nd month of the study to the end of the 6th month, the patient will be asked to do the Progressive Relaxation Exercise on their own for 30 minutes 3 days a week (Monday, Wednesday, Friday). No intervention will be made to the control group.
  Interventions: Other: sleep hygiene education and progressive relaxation exercise
- No intervention (No Intervention): No intervention will be made to the control group. Only data collection tools will be filled. Data collection tools (Individual identification form, PUKI, BAI) will be filled in face to face at the beginning (0th week), 8th and 12th weeks and at the end of the 6th month. The glycemic control of the patients will be evaluated with HbA1c checked every 3 months. Therefore, the HbA1c levels of the participants will be measured in the 0th and 12th weeks of the study and recorded on the follow-up form.

INTERVENTIONS:
Other: sleep hygiene education and progressive relaxation exercise — The study will be conducted with diabetic individuals who come to the endocrine clinic. The study will be conducted for 6 months. Intervention group Individuals who accept the study will be given face-to-face Progressive Relaxation Exercise training by the researcher in the first week of the first month of the study and will be applied. The Progressive Relaxation Exercise application will also be sent to the patient via WhatsApp and will be applied with the researcher via online interviews in the 2nd, 3rd and 4th weeks for 30 minutes 3 days a week (Monday-Wednesday-Friday). From the 2nd month of the study to the end of the 6th month, the patient will be asked to do the Progressive Relaxation Exercise on their own for 30 minutes 3 days a week (Monday, Wednesday, Friday). No intervention will be made to the control group.
  Arms: Experimental: intervention group

SUMMARY:
In diabetic patients, effective glycemic control is important in preventing complications, mortality and morbidity. The main purpose of DM treatment is to prevent neuropathic and vascular complications and to increase quality of life by keeping blood glucose levels and insulin activity within normal limits. It is stated that achieving the targeted glycemic control in diabetic patients reduces the risk of developing vascular complications in patients. In these patients, helping them reach the targeted glycemic level with lifestyle changes or medications is important in preventing the effects of diabetes on individual and community health. In effective DM monitoring and treatment, medical nutrition therapy (MNT), physical activity, drug therapy (OAD and insulin), DM education, patient self-monitoring and ensuring compliance with treatment are important. Although there have been significant developments in the field of treatment and follow-up today, there may be difficulties in achieving the targeted treatment goals in diabetic patients. This situation has led to the investigation of modifiable and non-modifiable factors affecting glycemic control in diabetic patients. Especially in Type 2 Diabetes, if these modifiable factors are diagnosed and managed early, effective management and control of diabetes can be achieved to a great extent. Especially psychological health and sleep health have become one of the new and mandatory modifiable risk factors for glycemic control in DM patients. Although it is known that diabetes is basically a disorder of the endocrine system, it has also been revealed that there is a relationship between psychosocial health and diabetes. Especially the presence of anxiety can cause an increase in blood glucose in diabetic patients, further worsening the patient's condition.Because emotional tension affects both neuroendocrine and hormonal pathways and indirectly the treatment and monitoring of diabetes, leading to blood sugar disorders. It is known that epinephrine secretion is stimulated by anxiety, which reduces the effect of insulin. Even in the simplest psychosocial stress and spiritual conflict, free fatty acids, cortisol and blood sugar increase. Therefore, stress and anxiety are considered important factors in patients whose blood sugar cannot be regulated despite medical treatment. In such cases, psychosocial evaluation should be made before increasing the insulin dose. In addition, studies in the literature show that in addition to the effect of anxiety on glycemic control, poor glycemic control also has an effect on the emergence of anxiety and a positive mutual relationship has been found between anxiety and glycemic control. Therefore, it was emphasized that anxiety and depression levels should be determined in order to consider diabetic patients as a whole. Sleep is a biological requirement and a physiologically active process. It repairs the body by giving strength to the mind and memory. Sleep quality is defined as the efficiency of sleep. Within the scope of sleep quality; sleep efficiency, number of sleep interruptions, total sleep duration, wakefulness duration, sleep transition time and spontaneous awakenings. Sleep, in addition to productivity and efficiency, positively affects cognitive functions such as memory and concentration, and contributes to physical and psychological renewal. Due to such positive effects, sleep is seen as an important variable affecting the individual's quality of life and well-being. Therefore, disruptions that may occur in sleep quality and sleep patterns cause problems such as inability to concentrate, anxiety, depression, increased sensitivity to pain, irritability, hallucinations, loss of appetite and difficulty in excretion, and directly affect the individual's daily life and general health. Therefore, it is important to take sleep health into consideration in order to ensure glycemic control in DM patients.

PURPOSE: This study will be conducted to examine the Effect of Sleep Hygiene Education and Progressive Relaxation Exercise on Sleep Quality, Anxiety and Glycemic Control in Type 2 Diabetic Patients.

DETAILED DESCRIPTION:
Today, it is known that sleep disorders are quite common in DM patients. In addition, it has been demonstrated that there is a two-way relationship between DM and sleep. The American Diabetes Association (ADA) included sleep as a behavior to be monitored among adults living with DM in its 2022 care standards .The American Academy of Sleep Medicine has also reported a relationship between sleep deprivation and sleep disorders and the progression or seriousness of DM, and stated that DM alone has an effect on sleep quality. Studies in the literature have also shown that sleep quality problems negatively affect diabetes, and a positive relationship has been found between poor sleep quality and hemoglobin A1c (HbA1c). The reason for this is; physiopathologically, in the NREM deep phase of sleep, sympathetic nerve activity decreases and the level of anti-insulin growth hormone increases, and in the second half of sleep, especially in the REM phase of sleep, the level of plasma cortisol, one of the anti-insulin regulatory hormones, increases.

In individuals with poor sleep quality and sleep disorders, the physiological state begins to deteriorate and glucose utilization decreases as a result of increased sympathetic activity, decreased growth hormone, and increased catecholamine and cortisol levels, and hyperglycemia and insulin resistance develop due to glycogenolysis and gluconeogenesis.Another reason is that short and poor sleep duration alters the ability of leptin, which has appetite suppressant properties, and ghrelin, which has appetite stimulant properties, to accurately report the body's calorie needs. This can lead to excessive calorie intake and obesity.Changes in the release of all these hormones that provide energy balance can lead to the risk of developing diabetes and deterioration in glycemic control and micro and macrovascular complications in people with diabetes. In the literature has been shown that insufficient sleep duration and decrease in sleep quality is associated with impaired glucose tolerance and insulin resistance. IAmong the reasons for this effect of sleep in these studies, it is stated that when sleep duration is insufficient and its quality is low, the risk of developing obesity, hyperglycemia and insulin resistance increases due to changes in the secretion of hormones that affect energy intake and expenditure. Therefore, it is important to consider sleep health in order to ensure glycemic control in DM patients. Nurses, who are in constant communication with patients, have important roles in determining the factors affecting the sleep quality of individuals and their sleep needs, diagnosing sleep disorders, and providing treatment. It is seen that the item "Sleep and rest", which is one of the physiological needs, is included in the nursing theory developed by Henderson, one of the important theorists. It is seen that the diagnosis of sleep pattern disturbance is also among the nursing diagnoses determined by NANDA. Therefore, sleep has an important role in nursing care. In addition, there are nursing interventions to improve sleep quality in DM patients. These interventions include sleep hygiene education, cognitive behavioral therapy, health education, music therapy, massage, aromatherapy. Among these interventions, in sleep hygiene education; not going to bed without feeling sleepy, not spending too much time in bed other than sleeping, not forcing yourself to fall asleep, setting sleep routines before going to bed, not taking daytime naps or sleeping, if taking daytime naps, not consuming carbonated drinks or caffeinated products at least 3-4 hours before going to bed, not going to bed hungry, avoiding heavy meals, stressful activities and strenuous movements before going to bed. Some studies were found that sleep hygiene training increased the quality of sleep in Type 2 DM patients. Relaxation exercises, which are effective in activating the parasympathetic system in DM patients, can also be used along with approaches such as sleep hygiene. Progressive relaxation exercise (PRE), one of these exercises, is a method that provides relaxation throughout the body by regularly and voluntarily relaxing large muscle groups in the human body. PRE is an intervention that nurses can teach. Relaxation exercises, one of the effective methods on anxiety and sleep; It is a widely used, effective and inexpensive method to change the behavior and mental processes of the individual. Recently, PGE has also started to be used in diabetes management. In an study conducted on diabetic patients, examining the effect of PGE on blood sugar, it was observed that there was a significant difference in the blood sugar levels of the experimental and control groups. The reason for this situation is thought to be due to the minimization of stress by controlling negative emotions with PGE . In another study examined the relationship between PGE and HbA1c in their randomized controlled study with Type 2 DM patients. According to the results of the study, positive improvements were observed in the HbA1c level of the experimental group, while there was no difference in the control group. It is thought that the reason for this situation is that hormonal activities become stable as PGE reduces stress Although the effects of PGE on sleep quality and glycemic control have been addressed separately in the literature, there is no study showing the effects on sleep quality and glycemic control at the same time. Therefore, it is thought that this study will emphasize the importance of using non-pharmacological interventions in the management of decreased sleep quality and anxiety affecting glycemic control in diabetic patients and will raise awareness about health professionals who apply these non-pharmacological interventions. In addition, it is thought that it will contribute to the literature because it is an evidence-based initiative in the field of nursing.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-65 years of age
* Literate
* Having a PSQI score >5
* Having been diagnosed with Type 2 diabetes for at least one year
* Having a mobile phone belonging to the person to be able to apply PGE
* Being able to use WhatsApp
* Those with a smartphone

Exclusion Criteria:

* Alcohol, sleeping pills, Sedative drugs, etc. that may affect sleep. those who use
* Those with HbA1c values >7
* Those who work night shifts
* Those with sleep disorders
* Those who are pregnant
* Those who are receiving pharmacological/non-pharmacological treatment due to a sleep disorder diagnosis
* Those with a vision, speech or hearing related disease that may prevent the understanding of the information given and the application of PGE
* Those with a chronic disease that may affect the quality of sleep (such as cancer, COPD, asthma), Those with a neuro-psychiatric disorder (such as dementia, psychotic disorder, bipolar disorder)
* Those whose condition is unstable and who develop a serious complication (such as retinopathy, nephropathy, neuropathy, etc.)
* Those with a disability that will prevent them from doing Progressive Relaxation Exercise
* Those who have any health problems during the application process
* Those who are receiving other complementary and alternative treatments during the application process
* Those who cannot continue the study for any reason, who want to withdraw from the study of their own free will and whose compliance with the progressive relaxation exercise and sleep hygiene training rules is less than 3 days
* Those whose diet and treatment changes during the study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | 6 months
  Data will be collected regarding the sleep quality scale be made at the beginning (week 0), immediately after the intervention 2 months (week 8) and 3 months (week 12) and at the end of the 6th month.The Pittsburgh Sleep Quality Index was developed by Buysse et al. (1989) in 1989. The validity and reliability of this scale in our country was determined by Ağargün et al. (1996) in 1996. The Cronbach Alpha internal consistency coefficient of the scale is 0.80. The coefficient being between 0.60-0.80 indicates that the reliability level is good. The PSQI consists of a total of 24 questions that evaluate the sleep quality in the last month. 19 of them are self-report questions. PSQI evaluate sleep quality in the last month. High component score averages indicate that sleep disturbances related to that component have increased. The total score has a value between 0-21.A PSQI global score of more than 5 is an indication of poor sleep quality.
Beck Anxiety Inventory (BAI) | 6 months
  Data will be collected regarding the BAI be made at the beginning (week 0), immediately after the intervention 2 months (week 8) and 3 months (week 12) and at the end of the 6th month. is a self-assessment scale developed by Beck and colleagues (1988) and used to determine the frequency of anxiety symptoms experienced by individuals. Its Turkish validity and reliability studies were conducted by Ulusoy and colleagues (1993). It is a Likert-type scale with a total of 21 self-assessment sentences, scored between 0 and 3. A high total score indicates a high level of anxiety or its severity. According to the scores obtained from the BAI, the anxiety levels of patients are; 0-17 points indicate low, 18-24 points indicate moderate, and 25 and above indicate a high level of anxiety.
Progressive Relaxation Exercise and Sleep Hygiene Training Compliance Chart | 6 months
  This chart was created with 3 options to determine how often individuals apply progressive relaxation exercise and sleep hygiene rules. In the literature, it has been determined that the frequency of PGE application varies between 4-12 weeks. Since individuals will be asked to do PGE exercise 3 days a week in this study, those who do it less than 3 days will be excluded from the study.

SECONDARY OUTCOMES:
The HbA1c levels of the participants | the HbA1c levels of the participants will be measured at the 0th and 12th weeks of the study and at the end of the 6th month and recorded on the follow-up form
  The glycemic control of the patients will be evaluated with HbA1c, which is checked every 3 months. Therefore, the HbA1c levels of the participants will be measured at the 0th and 12th weeks of the study and at the end of the 6th month and recorded on the follow-up form.

IPD SHARING:
Plan to Share IPD: No
The research will be used for scientific purposes and your individual identity information will remain confidential and will not be shared with anyone.

REFERENCES:
- [Background] 1. Hood, M. M., Reutrakul, S., Crowley, S. J. (2014). Night Eating İn Patients With Type 2 Diabetes. Associations with Glycemic Control, Eating Patterns, Sleep, and Mood. Appetite,79, 91- 96. 2. Sakamoto R,. Yamakawa, T., Takahashi,K. Suzuki,J., Shinoda, M.M., Sakamaki,K. Association of usual sleep quality and glycemic control in type 2 diabetes in Japanese: A cross sectional study. Sleep and Food Registry in Kanagawa (SOREKA). PLoS One2018 Jan 24;13(1):e0191771. 3. Akca, D. ve Saritas, S. (2021). Tip 2 diyabetli hastalarda gözlenen semptomlar ile uyku kalitesi arasındaki ilişki. Annals of Medical Research , 26 (4), 0579-0583. https://annalsmedres.org/index.php/aomr/article/view/1243. 4. Avianti, N., Desmaniarti, Z., & Rumahorbo, H. (2016). Progressive muscle relaxation effectiveness of the blood sugar patients with type 2 diabetes. Open Journal of Nursing, 6(3), 248-254. 5. Lou, P., Qin, Y., Zhang, P., Chen, P., Zhang, L., Chang, G., Li, T., Qiao, C., Zhang, N. (2015). Association Of Sleep Quality and Quality Of Life İn Type 2 Diabetes Mellitus: A Cross-Sectional Study İn China. Diabetes research and clinical practice, 107(1), 69-76. 6. Biggers, A., Barton, I., Henkins, J., Kim, H., Perez, R., Ong, J.,Sharp,L.K., Gerber, B.S. (2023). Association Between Sleep Hygiene Practices Scale And Sleep Quality İn Black and Latinx Patients With Uncontrolled Type 2 Diabetes.Sleep Med X, 2;5:100066. 7. Jamini,T. (2024).Theeffect of sleep hygiene on sleep quality of people with type 2 diabetes mellitus. Jurnal EduHealth, 15(01), 61-68. Retrieved from https://ejournal.seaninstitute.or.id/index.php/healt/article/view/3734 8. Amanda,S. P. (2019). Progressive musclerelaxation in improving sleep quality. Journal of Health, 6(2), 90-9 9. Trimurthula, S.R, Perakam, S., Kondapalli, A (2020). The Effect of Jacobson's Progressive Muscle Relaxation Technique along with Structured Exercise Program on HbA1c in Type II Diabetes Mellitus Patients. International Journal of Health S
- Available data/document: Informed Consent Form: sleep quality — https://etikkurullar.gazi.edu.tr/Dosya/Formlar — This study will be conducted in a randomized controlled and statistician blinded prospective design. During the blinding phase of the statistician; after the individuals are recruited to the study, the individuals will not be informed about which group they are in; 1 (Group 2: Control group), 2 (Group 1: Experimental group), and a coding will be created with the numbers 1 (Group 2: Control group), 2 (Group 1: Experimental group). The intervention and control groups will be assigned with simple random randomization. The individuals will be assigned numbers and the intervention and control groups will be assigned using the random number table. The analysis of the coded data by the groups will be done by a statistician. The coded groups will be delivered to the researcher in a sealed envelope by the statistician. Which code will be taken as the experimental and control groups will be determined by drawing lots.